CLINICAL TRIAL: NCT02835144
Title: Randomised Monocentric Clinical Study for the Identification of Cognitive and Neuroanatomical Alterations and for the Evaluation of the Efficacy of a Psychotherapeutic Intervention in Individuals With Risky Consumption of Alcohol and/or Sedative Drugs Aged ≥ 65 Years
Brief Title: Substance Use in Elderly Individuals: Brain and Cognitive Correlates and the Effect of Psychotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel changes; insufficient resources to continue
Sponsor: Prof. Dr. med. Egemen Savaskan (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Egemen Savaskan, Prof. Dr. med., Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNVRKAS - 2016-00210
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Substance Use Disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIQAAM_therapy (Experimental): Individuals in this group will receive units from the TIQAAM treatment program
  Interventions: Other: TIQAAM_therapy
- active_control (Active Comparator): Individuals in this group will receive units of psychoeducation
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: TIQAAM_therapy — The treatment program consists of TIQAAM therapy blocks to three priority areas: promoting change and motivation, relapse prevention and relapse management, and promote resource and euthymic activities to increase the abstinence motivation. The TIQAAM is based on behavioral approaches as well as motivational interviewing of Miller and Rollnick.
  Arms: TIQAAM_therapy
Other: Psychoeducation — This intervention is a psychoeducation module pertaining to substance use disorders.
  Arms: active_control

SUMMARY:
The prevalence of addictive disorders in old age is increasing. Age specific and appropriate therapeutic concepts tailored to in-patients thus represent a promising approach for the future. The investigated therapeutic intervention is a "therapy program for integrated qualified acute treatment of alcohol and drug problems" (TIQAAM).

DETAILED DESCRIPTION:
The prevalence of addictive disorders in old age is increasing. Age specific and appropriate therapeutic concepts tailored to inpatients thus represent a promising approach for the future. The investigated therapeutic intervention is a "therapy program for integrated qualified acute treatment of alcohol and drug problems" (TIQAAM).

Subjects ≥ 65 years, in which according to the WHO ASSIST V3.0 a risky consumption of alcoholic beverages, or benzodiazepines / non-benzodiazepine hypnotics (zolpidem, zopiclone, zaleplon), or both, are examined before and after a psychotherapeutic intervention during their inpatient stay exists. The data collected in part 1 of the study pertain to social integration, the motivation to change, quality of life in old age, general psychiatric symptoms. The data collected in part 2 of the study pertain to brain structure and functions. Data from standard procedures will be correlated to the data above.These relate to psychiatric symptoms, past consumption behavior, cognitive abilities, perceived social support and risk appetite.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 65 or above with, according to WHO-ASSIST V3.0, a hazardous consumption of alcoholic beverages and / or benzodiazepines and / or non-benzodiazepine hypnotics (zolpidem, zopiclone, zaleplon)
* The subjects must be able to understand verbal and written information about the study flow and content and to give their written consent.
* The subjects must be able to understand and perform verbal and written tasks (cognitive tests / questionnaires)

Exclusion Criteria:

* Taking medication that could affect cognition outside of benzodiazepines and / or non-benzodiazepine hypnotics (zolpidem, zopiclone, zaleplon).
* Drug treatments with anxiolytics (benzodiazepines) as part of an ongoing drug-assisted detoxification
* Taking antidepressant medication
* Taking sleep-inducing substances (for example Dipiperon®, Trittico®, Valverde Sleep® or Valverde Entspannung®)
* Taking other anxiolytic active substances (for example, pregabalin, Opipramol). The use of medication is allowed to treat somatic diseases.
* Use of drugs or substance dependence. Except for alcohol, benzodiazepines and non-benzodiazepine hypnotics (zolpidem, zopiclone, zaleplon)
* Diseases which prevent the subject from giving consent for this study or which impair cooperation in the investigation.
* Severe and / or unstable physical illness: severe depression, severe mania, delirium, severe cognitive impairment (mini-mental status test < 20/30 points), dementia of the Alzheimer type or other dementias, multiple sclerosis, clinically manifest structural brain damage (eg cerebral hemorrhage, brain tumors, MRI findings by Schulthess clinic)
* Heavily impaired vision and eye diseases

Additional exclusion criteria for part 2 of the study:

* Pacemaker, implantable cardioverter defibrillator (ICD), neurostimulator, aneurysm clip, prosthetic heart valve, valve prosthesis, metal prosthesis
* Clips after surgery, metallic bone plates, artificial joints, metal fragments in the body, professional in the metal processing industry, non-removable piercing, ferruginous tattoo ink
* Pregnancy
* Claustrophobia
* Use of alcohol or other consciousness-altering substances within 24 hours prior to the MRI scan (exceptions: see "exclusion criteria")

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
change in the total score of the Hospital Anxiety and Depression Scale - German version (HADS-D) | 210 days

CONTACTS AND LOCATIONS:
Overall Officials: Egemen Savaskan, Prof. Dr. med., Principal Investigator — Klinik für Alterspsychiatrie
Locations (1):
- Gerontopsychiatrisches Zentrum Hegibach, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided